CLINICAL TRIAL: NCT06241209
Title: Hemianopsia Rehabilitation After Stroke or Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00134526
Record Dates: First submitted 2023-12-08; First posted 2024-02-05 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Hemianopsia; Visual Field Defect, Peripheral; Visual Impairment
MeSH Terms: conditions — Hemianopsia; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (online news) (No Intervention): Group 1 with an odd number year of birth will be asked to view 15 minutes of online news three days per week for 2 months. LIVE: Canadian News | Weather & Traffic - Latest Sports | Breaking News (globalnews.ca)
- Group 2 (PowerPoint program) (Active Comparator): Group 2 with an even number year of birth will be asked to view the 15-minute PowerPoint program three days per week for 2 months.
  Interventions: Other: PowerPoint program visual stimulation

INTERVENTIONS:
Other: PowerPoint program visual stimulation — Moving objects, food, money, and other targets will be presented in the remaining seeing, and hemianopic areas.
  Arms: Group 2 (PowerPoint program)

SUMMARY:
In patients with hemianopsia following stroke or brain injury, we will determine if stimulating the visual field with images from a PowerPoint slide set can increase the visual field.

DETAILED DESCRIPTION:
Purpose: To determine if a computer screen visual stimulation can improve peripheral field loss in patients with vision pathway brain injury.

Hypothesis: Visual stimulation helps patients with visual pathway brain injury recover peripheral vision.

Justification: i) Axonal sprouting or re-rerouting can occur after brain injury ii) In Canada stroke prevalence comprises almost 900,000 patients. (Canada.ca, Health 2022). It is estimated that half of stroke survivors have a visual field deficit. (Rowe et al, PLoS One. 2019).

There is clinical equipoise regarding the results of vision therapy with visual stimulation. Romano JG, et al. Journal of the Neurological Sciences. 2008 Oct 15;273(1-2):70-4. versus Horton JC. Disappointing results from Nova Vision's visual restoration therapy. British Journal of Ophthalmology. 2005

Objectives: To determine the effect size of visual recovery, if any with computer screen visual stimulation

Research Method/Procedures

The project is prospective. Patients undergoing visual field testing found to have a hemianopsia will be invited to participate in the study. Chart review will be conducted on Connect Care. The following information will be collected: Patient age, sex, hand dominance, location and extent of stroke, number of prior strokes, time since initial/last stroke, neurologic diagnosis of neglect, perimetric findings, hours of television viewing, hours of smart phone use, hours of playing video games, smoking history, hypertension, diabetes mellitus, and hyperlipidemia.

Group 1 with an odd number year of birth will be asked to view 15 minutes of online news three days per week for 2 months. LIVE: Canadian News | Weather & Traffic - Latest Sports | Breaking News (globalnews.ca)

Group 2 with an even number year of birth will be asked to view the 15-minute PowerPoint program three days per week for 2 months.

At the end of 2 months, the study groups will be asked to cross over for 2 months, and perimetry will be repeated at month 4 from study entry. If patients originally in Group 2 do not want to stop using the PowerPoint program, they will be allowed to drop out of the study.

A 24-degree Humphrey automated perimetry will be performed at study entry, month two and month four. The perimeter provides a visual field index (VFI) with scores ranging from zero (no perceived light) to 100 (normal).

PLAN FOR DATA ANALYSIS: For each patient, the VFI from both eyes will be averaged. The difference between the pre-intervention and post-intervention VFI's will be compared between the PowerPoint intervention versus observation groups after 2 months. The same analysis will be repeated after the cross-over.

ELIGIBILITY:
Inclusion Criteria:

All patients 18 years of age or older with a homonymous hemianopsia or quadrantopsia, who can provide informed consent, and communicate in English.

Exclusion Criteria:

* The flashing lights from thge automated perimeter and PowerPoint program can potentially trigger photic seizures. Therefore patients with light-induced seizures are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Visual Field Index on Humphrey perimetry | 2 months
  (100 is an intact field)

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Institute of Alberta, Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://edseling.com